CLINICAL TRIAL: NCT00895882
Title: A Phase II Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Different Regimens of MK7009 When Administered Concomitantly With Pegylated Interferon and Ribavirin in Treatment-Naive Patients With Chronic Genotype 1 Hepatitis C Virus Infection
Brief Title: Study to Evaluate Different Regimens of Vaniprevir (MK7009) for the Treatment of Chronic Genotype 1 Hepatitis C Virus Infection in Treatment-naive Patients (MK-7009-019)(WITHDRAWN)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7009-019; 2009_586
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Genotype 1 Hepatitis C Virus Infection
MeSH Terms: interventions — vaniprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): vaniprevir 300 mg b.i.d. + peg-IFN + RBV for 12 weeks, followed by placebo to vaniprevir + peg-IFN + RBV for 12 weeks
  Interventions: Drug: vaniprevir (MK7009); Drug: Comparator: Pegylated Interferon (peg-IFN) alfa-2a; Drug: Comparator: Ribavirin; Drug: Comparator: Placebo to vaniprevir
- 2 (Experimental): vaniprevir 300 mg b.i.d. + peg-IFN + RBV for 24 weeks
  Interventions: Drug: vaniprevir (MK7009); Drug: Comparator: Pegylated Interferon (peg-IFN) alfa-2a; Drug: Comparator: Ribavirin
- 3 (Experimental): vaniprevir 600 mg b.i.d. + peg-IFN + RBV for 12 weeks, followed by placebo to vaniprevir + peg-IFN + RBV for 12 weeks
  Interventions: Drug: Comparator: vaniprevir (MK7009); Drug: Comparator: Pegylated Interferon (peg-IFN) alfa-2a; Drug: Comparator: Ribavirin; Drug: Comparator: Placebo to vaniprevir
- 4 (Experimental): vaniprevir 600 mg b.i.d. + peg-IFN + RBV for 24 weeks
  Interventions: Drug: Comparator: vaniprevir (MK7009); Drug: Comparator: Pegylated Interferon (peg-IFN) alfa-2a; Drug: Comparator: Ribavirin
- 5 (Experimental): vaniprevir 600 mg q.d. + peg-IFN + RBV for 24 weeks
  Interventions: Drug: Comparator: vaniprevir (MK7009); Drug: Comparator: Pegylated Interferon (peg-IFN) alfa-2a; Drug: Comparator: Ribavirin
- 6 (Placebo Comparator): Placebo to vaniprevir + peg-IFN + RBV for 24 weeks, followed by peg-IFN + RBV for 24 weeks
  Interventions: Drug: Comparator: Pegylated Interferon (peg-IFN) alfa-2a; Drug: Comparator: Ribavirin; Drug: Comparator: Placebo to vaniprevir

INTERVENTIONS:
Drug: vaniprevir (MK7009) — vaniprevir 300 mg soft gel capsules twice daily.
  Arms: 1; 2
Drug: Comparator: vaniprevir (MK7009) — vaniprevir 600 mg soft gel capsules twice daily.
  Arms: 3; 4; 5
Drug: Comparator: Pegylated Interferon (peg-IFN) alfa-2a — Peg-IFN 180 mcg/0.5 mL subcutaneous injection once weekly
Drug: Comparator: Ribavirin — Ribavirin, at a total daily dose of 1000 mg or 1200 mg based on patient weight, will be administered twice daily.
Drug: Comparator: Placebo to vaniprevir — Placebo to vaniprevir soft gel capsules twice daily.
  Arms: 1; 3; 6

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of vaniprevir when administered concomitantly with pegylated interferon (peg-IFN) and ribavirin (RBV) to treat treatment-naive genotype 1 hepatitis C virus (HCV)-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic genotype 1 HCV infection
* Patient has had a liver biopsy without evidence of cirrhosis
* Patient has had an eye exam prior to the start of study
* Female patients capable of having children and male patients with female partners capable of having children agree to use two forms of birth control throughout the study

Exclusion Criteria:

* Patient has had previous treatment with: 3 or more doses IFN, peg-IFN, and/or RBV; and stopped treatment due to intolerance of one of the drugs; other antiviral or investigational therapies or vaccines for HCV
* Female patient is pregnant or breastfeeding
* Patient has chronic hepatitis not caused by HCV
* Patient has evidence of cirrhosis of the liver
* Patient has HIV
* Patient has active hepatitis B infection
* Patient has non-genotype 1 HCV infection
* Patient consumes excessive amounts of alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving SVR24 in Treatment Regimens 1 to 4 | 24 weeks after end of study therapy
Evaluate the safety and tolerability of the MK7009 treatment regiments as assessed by review of the accumulated safety data | 72 Weeks

SECONDARY OUTCOMES:
1) Proportion of patients achieving SVR24 in Treatment Regimen 5 | 1) 24 weeks after end of study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC